CLINICAL TRIAL: NCT06014853
Title: A Randomized, Open-label, Four-sequence, Four-period, Crossover, Single Dosing, Phase 1 Clinical Trial to Compare the Safety, Tolerability, and Pharmacokinetics of SOL-804 and Zytiga in Healthy Male Subjects
Brief Title: A Study to Evaluate Safety, Tolerability, and Pharmacokinetics of SOL-804 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Collaborators: Dyna Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DN-SOL-102
Record Dates: First submitted 2023-08-14; First posted 2023-08-28 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: Abiraterone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Period 1: Zytiga® 1000mg / Period 2 : SOL-804-F 302.5mg / Period 3 : SOL-804-F 242.0mg / Period 4 : SOL-804-F 181.5mg
  Interventions: Drug: SOL-804-F; Drug: Zytiga
- Group 2 (Experimental): Period 1 : SOL-804-F 181.5mg / Period 2 : Zytiga® 1000mg / Period 3 : SOL-804-F 302.5mg / Period 4 : SOL-804-F 242.0mg
  Interventions: Drug: SOL-804-F; Drug: Zytiga
- Group 3 (Experimental): Period 1 : SOL-804-F 242.0mg / Period 2 : SOL-804-F 181.5mg / Period 3 Zytiga® 1000mg / Period 4 : SOL-804-F 302.5mg
  Interventions: Drug: SOL-804-F; Drug: Zytiga
- Group 4 (Experimental): Period 1 : SOL-804-F 302.5mg / Period 2 : SOL-804-F 242.0mg / Period 3 : SOL-804-F 181.5mg / Period 4 : Zytiga® 1000mg
  Interventions: Drug: SOL-804-F; Drug: Zytiga

INTERVENTIONS:
Drug: SOL-804-F — All subjects who have been fasting for at least 10 hours prior to administration will take investigational products orally with water on the administration day of each period.
  Other Names: SOL-804-F 181.5mg/242.0mg/302.5mg
Drug: Zytiga — All subjects who have been fasting for at least 10 hours prior to administration will take investigational products orally with water on the administration day of each period.
  Other Names: Zytiga 500mg

SUMMARY:
Study Design : A randomized, open-label, four-sequence, four-period, crossover, single dosing, phase 1 study

DETAILED DESCRIPTION:
To evaluate the safety, tolerability and pharmacokinetic characteristics of SOL-804-F and Zytiga tablets following a single oral dose and Zytiga 1,000 mg in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. healthy adult male volunteers between 19 to 50 years of age at screening visit.
2. Body mass index (BMI) between 19.0 to 30.0 kg/m2
3. The subjects voluntarily decide to participate in the study after receiving a full explanation and understanding and provide written consent
4. The subjects are suitable for this study as determined by the investigator (physical examination, clinical laboratory tests, etc.)

Exclusion Criteria:

1. Clinically significant abnormal physical examination, vital signs or ECG
2. The subjects who have a medical history of hepatobiliary, renal, neurological, immune, respiratory, endocrine, hematologic, oncologic, cardiovascular, urinary, psychiatric or sexual dysfunction.
3. The subjects who have a hereditary disorder including galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption, etc.
4. The subjects who have a history of drug abuse or positive with urine drug screening test

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
AUClast of abiraterone | 72 hours
  Area under the plasma drug concentration-time curve from 0 to last
Cmax of abiraterone | 72 hours
  The maximum or peak concentration between zero and dosing interval

SECONDARY OUTCOMES:
AUCinf of abiraterone | 72 hours
  Area under the plasma drug concentration-time curve from 0 to infinity
Tmax of abiraterone | 72 hours
  Time of Maximum Concentration
t1/2 of abiraterone | 72 hours
  Terminal Half-life
CL/F of abiraterone | 72 hours
  An estimate of the total body clearance after oral administration
Vd/F of abiraterone | 72 hours
  Apparent volume of distribution after extravascular administration

OTHER OUTCOMES:
Rmax of serum testosterone | 72 hours
  The maximum response
Imax of serum testosterone | 72 hours
  Maximum inhibition

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No